CLINICAL TRIAL: NCT07176234
Title: Linking Exericise for Advancing Daily Stress (LEADS) Management and Resilience in African American Families
Brief Title: The LEADS Trial (Linking Exericise for Advancing Daily Stress Management)
Acronym: LEADS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Dawn Wilson, Professor of Psychology, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00135549; R01MD019714 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-01

CONDITIONS: Obesity, Childhood
Keywords: physical activity, stress management, adolescent, intervention, African American
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized group cohort study design
Who Masked: Outcomes Assessor
Masking Description: All measurement staff are blind to conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Health Education (Active Comparator): Includes a series of health education sessions, including hypertension, diabetes, cancer, sleep, social media advocacy, metabolism, financial literacy.
  Interventions: Other: Health Education
- Intervention Arm (Experimental): Behavioral Intervention for reducing stress and increasing resilience for improve physical activity, healthy diet, and wellbeing
  Interventions: Behavioral: Treatment

INTERVENTIONS:
Behavioral: Treatment — The Linking Exercise for Advancing Daily Stress (LEADS) Management intervention integrates a family-based intervention to address chronic stressors to promote behavioral skills for increasing PA in overweight AA adolescents and their parents. Based on Lazarus and Folkman's Stress and Coping Model, Family Systems, and Social Cognitive Theories, the proposed intervention integrates components that build coping skills (mindfulness, deep breathing, active coping, cognitive reframing), self-esteem (self-affirmation), and positive parenting practices (parent support, nurturance, family routines).
  Arms: Intervention Arm
Other: Health Education — Attention Control Comparator
  Arms: Comprehensive Health Education

SUMMARY:
Chronic stressors have wide-reaching harmful effects on the physical, social, and psychological well-being of many African American (AA) families. These stressors place some AA adolescents, who already experience low rates of physical activity (PA) and high rates of obesity, at even greater risk for developing chronic diseases. Previous family-based interventions have targeted PA, diet, and sedentary behaviors to prevent and manage overweight and obesity, but few have been successful for AA adolescents. The investigators propose that this may be because chronic stressors are a major challenge to engagement in health promotion efforts, which has been significantly overlooked in previous interventions for AA families. Resilience-based interventions that empower youth to cope with daily stressors have shown improvements across a broad range of outcomes including mental health, academic achievement, and risk-taking behaviors. However, no previous study has evaluated a family-based stress and coping plus positive parenting intervention on improving engagement in PA in AA families. The Linking Exercise for Advancing Daily Stress (LEADS) Management intervention integrates a family-based intervention to address chronic stressors to promote behavioral skills for increasing PA in overweight AA adolescents and their parents. Based on Lazarus and Folkman's Stress and Coping Model, Family Systems, and Social Cognitive Theories, the proposed intervention integrates components that build coping skills (mindfulness, deep breathing, active coping, cognitive reframing), self-esteem (self-affirmation), and positive parenting practices (parent support, nurturance, family routines). The investigators propose that these protective factors as integrated into the LEADS intervention will buffer the negative effects of chronic stressors, which will lead to greater improvements in PA. The investigators pilot research indicates that the LEADS family-based intervention was feasible and acceptable and led to increased moderate-to-vigorous PA (MVPA) for adolescents. Thus, the primary aim of this study is 1) to evaluate the efficacy of the LEADS intervention on increasing MVPA from baseline to post-intervention, and maintenance at a 6-month follow-up in overweight AA adolescents. Secondary aims will examine 2) the effect of the LEADS intervention on light PA, dietary intake, family mealtime, body mass index, waist circumference, and blood pressure outcomes, 3) the effects of the intervention on parent outcomes, as well as examining 4) mediators of the intervention effect on changes in PA.

ELIGIBILITY:
Inclusion Criteria:

* adolescent BMI greater than or equal 70th percentile;
* self-identified African American or Black adolescents 11-16 years;
* at least one parent/caregiver participating;
* not currently in a structured physical activity, weight loss program or stress management program
* access to the internet in his/her home.

Exclusion Criteria:

* having limitations that would prevent physical activity, and for caregivers,
* criteria will include having a cardiovascular or orthopedic condition that would limit physical activity
* uncontrolled blood pressure.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2029-08-10 (Estimated); Study Completion 2029-08-10 (Estimated)

PRIMARY OUTCOMES:
daily minutes of moderate to vigorous physical activity | baseline, post-10 week group session, 6-month follow-up
  7-day accelerometer estimates using actigraph

SECONDARY OUTCOMES:
daily minuties of light physical activity | baseline, post-10 week group session, 6-month follow up
  7-day accelerometer estimates using actigraph
body mass index | baseline, post-10 week group session, 6 month follow-up
  weight (kg)/ height (m)2
Adolescent Self-Regulation | baseline, post 10 week group session, 6 month follow up
  Self-Regulation self report scale ranging from 7-35 (higher values are more positive)
Wellbeing | baseline, post 10 week group session, 6 month follow up
  Psychological wellbeing scale ranging from 24-120 (with higher values being more positive)
Coping with Stress | Baseline, post 10 week group session, 6 month follow up
  Brief Cope Scale is a self report scale ranging from 10-40 (with higher scores being more positive)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - M.H. Newton Family Life Enrichment Center, Sumter, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from 330 Black/African American families (parent/adolescent dyads). We will make available behavioral, psychosocial, physiological, and physical activity data after the data provided by this grant has been published in peer-reviewed journals, consistent with the Final NIH Statement on Sharing Research Data. The final dataset will be stripped of identifiers prior to release for sharing. Data will be made available in a format consistent with community standards in a spreadsheet-based data exchange format. Once available, data can be requested by email to the Principal Scientific Investigator. Regarding our management of intellectual property, we will adhere to the NIH Policy on Sharing of Unique Research Resources as specified in Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the trial has been completed and published we will make the data available.
Access Criteria: Data Preservation, Access, and Associated Timeline The study data will be submitted to a repository that is participating in the NIH Generalist Repository Initiative. We will submit metadata associated with the datasets to Vivli. Scientific data will be shared as soon as possible.
  Access, Distribution and Reuse The study datasets will be collected following informed consent as set by the NIH and IRB at the University of South Carolina. To protect research participants' privacy and confidentiality, data submitted to the repository will not include personal identifiable information such as names or addresses.